CLINICAL TRIAL: NCT00048958
Title: Cytogenetic Studies in Acute Leukemia and Multiple Myeloma: Companion to CALGB Treatment Studies For Previously Untreated Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), Myelodysplastic Syndrome (MDS) or Multiple Myeloma (MM) Patients
Brief Title: Cytogenetic Studies in Acute Leukemia and Multiple Myeloma
Status: Active, not recruiting | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-8461; NCI-2009-00494 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); CDR0000256897 (Registry Identifier: PDQ (Physician Data Query)); 3U24CA114725-09S1 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Multiple Myeloma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Multiple Myeloma | interventions — Cytogenetic Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Institutions must submit patient samples (eg, bone marrow and peripheral blood) at diagnosis, at complete remission, and at the time of relapse to the Alliance-Approved Institutional Cytogeneticist.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Samples as defined per the protocol for previously untreated patients with AML, ALL, MDS or MM will be submitted for analysis and within one month patients are required to register onto a CALGB treatment study.
  Interventions: Genetic: cytogenetic analysis

INTERVENTIONS:
Genetic: cytogenetic analysis

SUMMARY:
Chromosomal analysis or the study of genetic differences in patients previously untreated with AML, ALL, MDS or MM may be helpful in the diagnosis and classification of disease. It may also improve the ability to predict the course of disease and the selection of therapy. Institutions must have either an Alliance-approved cytogeneticist or an agreement from an Alliance-approved main member cytogenetics laboratory to enroll a patient on CALGB 8461. The Alliance Approved Institutional Cytogeneticists list is posted on the Alliance for Clinical Trials in Oncology website.

ELIGIBILITY:
1. Patients from adjuncts are eligible if the Main Member Cytogenetics laboratory has agreed to process samples from that adjunct.
2. Within one month of registration on CALGB 8461, register onto a CALGB treatment study for previously untreated AML, ALL, MDS, or MM patients.
3. Simultaneously with registration on CALGB 8461, register patients within the continental United States onto CALGB 9665 (LTB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population from the clinical oncology research community including academic institutions, hospitals and clinics.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 1984-06 (Actual); Primary Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of specific less common primary as well as common secondary chromosome abnormalities in adult AML, ALL, MDS and MM | Up to 10 years
Correlate specific (normal or various primary and secondary chromosomal abnormalities) with clinical and laboratory parameters | Up to 10 years
Correlate specific karyotype groups with response rates, response duration, survival and cure in patients treated with various induction and post-induction regimens | Up to 10 years
Correlate specific karyotype groups with selected molecular abnormalities as studied in CALGB leukemia protocols | Up to 10 years
To correlate specific karyotype groups with multidrug resistance data | Up to 10 years
To correlate specific karyotype groups with epidemiologic data (toxic exposure and family history) | Up to 10 years
To determine karyotype changes at relapse and the influence of the type of change (or no change) in karyotype at relapse on subsequent clinical course | up to 10 yeras
To identify new chromosome abnormalities important in leukemogenesis | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bloomfield, MD, Study Chair — James Cancer Hospital and Solove Research Institute
Locations (137):
- United States (137):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Marcucci G, Mrozek K, Ruppert AS, Maharry K, Kolitz JE, Moore JO, Mayer RJ, Pettenati MJ, Powell BL, Edwards CG, Sterling LJ, Vardiman JW, Schiffer CA, Carroll AJ, Larson RA, Bloomfield CD. Prognostic factors and outcome of core binding factor acute myeloid leukemia patients with t(8;21) differ from those of patients with inv(16): a Cancer and Leukemia Group B study. J Clin Oncol. 2005 Aug 20;23(24):5705-17. doi: 10.1200/JCO.2005.15.610. PMID 16110030
- [Background] Mrozek K, Carroll AJ, Maharry K, et al.: Central review of cytogenetics is essential for cooperative group clinical and correlative studies of acute leukemia: The Cancer and Leukemia Group B (CALGB) 8461 experience. [Abstract] Blood 104 (11): A-1081, 2004.
- [Background] Sekeres MA, Peterson B, Dodge RK, Mayer RJ, Moore JO, Lee EJ, Kolitz J, Baer MR, Schiffer CA, Carroll AJ, Vardiman JW, Davey FR, Bloomfield CD, Larson RA, Stone RM; Cancer and Leukemia Group B. Differences in prognostic factors and outcomes in African Americans and whites with acute myeloid leukemia. Blood. 2004 Jun 1;103(11):4036-42. doi: 10.1182/blood-2003-09-3118. Epub 2004 Feb 19. PMID 14976037
- [Background] Baldus CD, Tanner SM, Ruppert AS, Whitman SP, Archer KJ, Marcucci G, Caligiuri MA, Carroll AJ, Vardiman JW, Powell BL, Allen SL, Moore JO, Larson RA, Kolitz JE, de la Chapelle A, Bloomfield CD. BAALC expression predicts clinical outcome of de novo acute myeloid leukemia patients with normal cytogenetics: a Cancer and Leukemia Group B Study. Blood. 2003 Sep 1;102(5):1613-8. doi: 10.1182/blood-2003-02-0359. Epub 2003 May 15. PMID 12750167
- [Background] Heinonen K, Rao PN, Slack JL, Cruz J, Bloomfield CD, Mrozek K. Isochromosome 12p in two cases of acute myeloid leukaemia without evidence of germ cell tumour. Br J Haematol. 1996 Jun;93(3):677-80. doi: 10.1046/j.1365-2141.1996.d01-1687.x. PMID 8652392
- [Result] Cancer and Leukemia Group B 8461; Farag SS, Archer KJ, Mrozek K, Ruppert AS, Carroll AJ, Vardiman JW, Pettenati MJ, Baer MR, Qumsiyeh MB, Koduru PR, Ning Y, Mayer RJ, Stone RM, Larson RA, Bloomfield CD. Pretreatment cytogenetics add to other prognostic factors predicting complete remission and long-term outcome in patients 60 years of age or older with acute myeloid leukemia: results from Cancer and Leukemia Group B 8461. Blood. 2006 Jul 1;108(1):63-73. doi: 10.1182/blood-2005-11-4354. Epub 2006 Mar 7. PMID 16522815
- [Result] Farag SS, Ruppert AS, Mrozek K, Mayer RJ, Stone RM, Carroll AJ, Powell BL, Moore JO, Pettenati MJ, Koduru PR, Stamberg J, Baer MR, Block AW, Vardiman JW, Kolitz JE, Schiffer CA, Larson RA, Bloomfield CD. Outcome of induction and postremission therapy in younger adults with acute myeloid leukemia with normal karyotype: a cancer and leukemia group B study. J Clin Oncol. 2005 Jan 20;23(3):482-93. doi: 10.1200/JCO.2005.06.090. Epub 2004 Nov 8. PMID 15534356
- [Result] Bloomfield CD, Ruppert AS, Mrozek K, Kolitz JE, Moore JO, Mayer RJ, Edwards CG, Sterling LJ, Vardiman JW, Carroll AJ, Pettenati MJ, Stamberg J, Byrd JC, Marcucci G, Larson RA; Cancer and Leukemia Group B (CALGB) Study 8461. Core binding factor acute myeloid leukemia. Cancer and Leukemia Group B (CALGB) Study 8461. Ann Hematol. 2004;83 Suppl 1:S84-5. doi: 10.1007/s00277-004-0850-2. No abstract available. PMID 15124687
- [Result] Blum W, Mrozek K, Ruppert AS, et al.: Early allogeneic transplantation for adults with de novo acute myeloid leukemia presenting with t(6;11)(q27;q23): results from CALGB 8461. [Abstract] J Clin Oncol 22 (Suppl 14): A-6543, 568s, 2004.
- [Result] Blum W, Mrozek K, Ruppert AS, Carroll AJ, Rao KW, Pettenati MJ, Anastasi J, Larson RA, Bloomfield CD. Adult de novo acute myeloid leukemia with t(6;11)(q27;q23): results from Cancer and Leukemia Group B Study 8461 and review of the literature. Cancer. 2004 Sep 15;101(6):1420-7. doi: 10.1002/cncr.20489. PMID 15368330
- [Result] Byrd JC, Ruppert AS, Mrozek K, Carroll AJ, Edwards CG, Arthur DC, Pettenati MJ, Stamberg J, Koduru PR, Moore JO, Mayer RJ, Davey FR, Larson RA, Bloomfield CD. Repetitive cycles of high-dose cytarabine benefit patients with acute myeloid leukemia and inv(16)(p13q22) or t(16;16)(p13;q22): results from CALGB 8461. J Clin Oncol. 2004 Mar 15;22(6):1087-94. doi: 10.1200/JCO.2004.07.012. PMID 15020610
- [Result] Farag SS, Archer KJ, Mrózek K, et al.: Pre-treatment cytogenetics predict complete remission and long-term outcome in patients (Pts) ≥60 years with acute myeloid leukemia (AML): results from Cancer and Leukemia Group B (CALGB) 8461. [Abstract] Blood 104 (11): A-568, 2004.
- [Result] Marcucci G, Mrózek, K, Ruppert AS, et al.: t(8;21) Acute myeloid leukemia (AML) differs from inv(16) AML in pretreatment characteristics, outcome and prognostic factors predicting outcome: a Cancer and Leukemia Group B (CALGB) Study. [Abstract] Blood 104 (11): A-2017, 2004.
- [Result] Marcucci G, Mrozek K, Ruppert AS, Archer KJ, Pettenati MJ, Heerema NA, Carroll AJ, Koduru PR, Kolitz JE, Sterling LJ, Edwards CG, Anastasi J, Larson RA, Bloomfield CD. Abnormal cytogenetics at date of morphologic complete remission predicts short overall and disease-free survival, and higher relapse rate in adult acute myeloid leukemia: results from cancer and leukemia group B study 8461. J Clin Oncol. 2004 Jun 15;22(12):2410-8. doi: 10.1200/JCO.2004.03.023. PMID 15197203
- [Result] Slovak ML, Bloomfield CD, Gundacker H, et al.: Acute myeloid leukemia (AML) with t(6;9)(p23;q34) defines a very poor risk leukemia subgroup with distinguishing clinicopathological features: a United States (US) Cytogenetics Intergroup Study of 62 AML and MDS cases. [Abstract] Blood 104 (11): A-567, 2004.
- [Result] Byrd JC, Mrozek K, Dodge RK, Carroll AJ, Edwards CG, Arthur DC, Pettenati MJ, Patil SR, Rao KW, Watson MS, Koduru PR, Moore JO, Stone RM, Mayer RJ, Feldman EJ, Davey FR, Schiffer CA, Larson RA, Bloomfield CD; Cancer and Leukemia Group B (CALGB 8461). Pretreatment cytogenetic abnormalities are predictive of induction success, cumulative incidence of relapse, and overall survival in adult patients with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B (CALGB 8461). Blood. 2002 Dec 15;100(13):4325-36. doi: 10.1182/blood-2002-03-0772. Epub 2002 Aug 1. PMID 12393746
- [Result] Farag SS, Archer KJ, Mrozek K, Vardiman JW, Carroll AJ, Pettenati MJ, Moore JO, Kolitz JE, Mayer RJ, Stone RM, Larson RA, Bloomfield CD. Isolated trisomy of chromosomes 8, 11, 13 and 21 is an adverse prognostic factor in adults with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B 8461. Int J Oncol. 2002 Nov;21(5):1041-51. PMID 12370753
- [Result] Bloomfield CD, Byrd JC, Farag SS, et al.: Cytogenetics for treatment stratification in adult acute myeloid leukemia (AML). [Abstract] Ann Hematol 80 (Suppl 2): A-37, S10, 2001.
- [Result] Farag SS, Archer KJ, Carroll AJ, et al.: Isolated trisomy (IT) is an adverse prognostic factor in patients (pts) with AML: results from Cancer and Leukemia Group B (CALGB 8461). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1124, 2001.
- [Result] Marcucci G, Archer KJ, Mrózek K, et al.: Abnormal karyotype during complete remission (CR) predicts short relapse-free survival (RFS) in acute myeloid leukemia (AML): results from CALGB 8461. [Abstract] Blood 98 (11 Pt 1): A-2421, 577a, 2001.
- [Result] Wetzler M, Dodge RK, Mrozek K, et al.: Secondary chromosome aberrations in adult acute lymphoblastic leukemia (ALL) with t(9;22) - a Cancer and Leukemia Group B (CALGB) study. [Abstract] Blood 98 (11 Pt 1): A-466, 111a, 2001.
- [Result] Wetzler M, Dodge RK, Mrózek K, et al.: Karyotype change in adult acute myeloid leukemia (AML) at first relapse - CALGB 8461. [Abstract] Blood 96 (11 Pt 1): A-3046, 706a, 2000.
- [Result] Bloomfield D: Adult acute myeloid leukemia (AML) patients (PTS) with t(8;21)(q22;q22) have a superior outcome when repetitive cycles of high-dose cytarabine (HDAC) are administered. [Abstract] Ann Hematol 78 (Suppl 2): A-50, S13, 1999.
- [Result] Byrd JC, Dodge RK, Carroll A, Baer MR, Edwards C, Stamberg J, Qumsiyeh M, Moore JO, Mayer RJ, Davey F, Schiffer CA, Bloomfield CD. Patients with t(8;21)(q22;q22) and acute myeloid leukemia have superior failure-free and overall survival when repetitive cycles of high-dose cytarabine are administered. J Clin Oncol. 1999 Dec;17(12):3767-75. doi: 10.1200/JCO.1999.17.12.3767. PMID 10577848
- [Result] Wetzler M, Dodge RK, Mrozek K, Carroll AJ, Tantravahi R, Block AW, Pettenati MJ, Le Beau MM, Frankel SR, Stewart CC, Szatrowski TP, Schiffer CA, Larson RA, Bloomfield CD. Prospective karyotype analysis in adult acute lymphoblastic leukemia: the cancer and leukemia Group B experience. Blood. 1999 Jun 1;93(11):3983-93. PMID 10339508
- [Result] Baer MR, Stewart CC, Lawrence D, Arthur DC, Mrozek K, Strout MP, Davey FR, Schiffer CA, Bloomfield CD. Acute myeloid leukemia with 11q23 translocations: myelomonocytic immunophenotype by multiparameter flow cytometry. Leukemia. 1998 Mar;12(3):317-25. doi: 10.1038/sj.leu.2400933. PMID 9529125
- [Result] Bloomfield CD, Lawrence D, Byrd JC, Carroll A, Pettenati MJ, Tantravahi R, Patil SR, Davey FR, Berg DT, Schiffer CA, Arthur DC, Mayer RJ. Frequency of prolonged remission duration after high-dose cytarabine intensification in acute myeloid leukemia varies by cytogenetic subtype. Cancer Res. 1998 Sep 15;58(18):4173-9. PMID 9751631
- [Result] Byrd JC, Dodge R, Carroll A, et al.: Adult acute myeloid leukemia (AML) patients (PTS) with t(8;21)(q22;q22) have a superior outcome when repetitive cycles of high-dose cytarabine (HDAC) are administered. [Abstract] Blood 92 (10 Pt 1): A-1282, 312a, 1998.
- [Result] Byrd JC, Lawrence D, Arthur DC, Pettenati MJ, Tantravahi R, Qumsiyeh M, Stamberg J, Davey FR, Schiffer CA, Bloomfield CD. Patients with isolated trisomy 8 in acute myeloid leukemia are not cured with cytarabine-based chemotherapy: results from Cancer and Leukemia Group B 8461. Clin Cancer Res. 1998 May;4(5):1235-41. PMID 9607582
- [Result] Caligiuri MA, Strout MP, Lawrence D, Arthur DC, Baer MR, Yu F, Knuutila S, Mrozek K, Oberkircher AR, Marcucci G, de la Chapelle A, Elonen E, Block AW, Rao PN, Herzig GP, Powell BL, Ruutu T, Schiffer CA, Bloomfield CD. Rearrangement of ALL1 (MLL) in acute myeloid leukemia with normal cytogenetics. Cancer Res. 1998 Jan 1;58(1):55-9. PMID 9426057
- [Result] Heinonen K, Mrozek K, Lawrence D, Arthur DC, Pettenati MJ, Stamberg J, Qumsiyeh MB, Verma RS, MacCallum J, Schiffer CA, Bloomfield CD. Clinical characteristics of patients with de novo acute myeloid leukaemia and isolated trisomy 11: a Cancer and Leukemia Group B study. Br J Haematol. 1998 Jun;101(3):513-20. doi: 10.1046/j.1365-2141.1998.00714.x. PMID 9633896
- [Result] Wetzler M, Dodge RK, Mrózek K, et al.: Trisomy 8 represents a poor risk group in adult acute lymphoblastic leukemia (ALL): results from Cancer and Leukemia Group B (CALGB) 8461. [Abstract] Blood 92 (10 Pt 1): A-914, 223a, 1998.
- [Result] Byrd JC, Weiss RB, Arthur DC, Lawrence D, Baer MR, Davey F, Trikha ES, Carroll AJ, Tantravahi R, Qumsiyeh M, Patil SR, Moore JO, Mayer RJ, Schiffer CA, Bloomfield CD. Extramedullary leukemia adversely affects hematologic complete remission rate and overall survival in patients with t(8;21)(q22;q22): results from Cancer and Leukemia Group B 8461. J Clin Oncol. 1997 Feb;15(2):466-75. doi: 10.1200/JCO.1997.15.2.466. PMID 9053467
- [Result] Mrózek K, Heinonen K, Lawrence D, et al.: t(9;11)(p22;q23) confers better prognosis than other translocations of 11q23 in adults with de novo acute myeloid leukemia (AML): a Cancer and Leukemia Group B study. [Abstract] Cytogenet Cell Genet 77: A-P332, 136, 1997.
- [Result] Mrozek K, Heinonen K, Lawrence D, Carroll AJ, Koduru PR, Rao KW, Strout MP, Hutchison RE, Moore JO, Mayer RJ, Schiffer CA, Bloomfield CD. Adult patients with de novo acute myeloid leukemia and t(9; 11)(p22; q23) have a superior outcome to patients with other translocations involving band 11q23: a cancer and leukemia group B study. Blood. 1997 Dec 1;90(11):4532-8. PMID 9373264
- [Result] Bernstein SH, Brunetto VL, Davey FR, Wurster-Hill D, Mayer RJ, Stone RM, Schiffer CA, Bloomfield CD. Acute myeloid leukemia-type chemotherapy for newly diagnosed patients without antecedent cytopenias having myelodysplastic syndrome as defined by French-American-British criteria: a Cancer and Leukemia Group B Study. J Clin Oncol. 1996 Sep;14(9):2486-94. doi: 10.1200/JCO.1996.14.9.2486. PMID 8823327
- [Result] Byrd JC, Lawrence D, Arthur DC, et al.: Acute myeloid leukemia (AML) patients with pre-treatment isolated trisomy 8 are rarely cured with chemotherapy: results of CALGB 8461. [Abstract] Proc Am Assoc Cancer Res 37: A-1286, 188, 1996.
- [Result] Caligiuri MA, Strout MP, Arthur DC, et al.: Rearrangement of ALL1 is a recurrent molecular defect in adult acute myeloid leukemia (AML) with normal cytogenetics that predicts a short complete remission (CR) duration. [Abstract] Proceedings of the American Society of Clinical Oncology 15: A-1060, 1996.
- [Result] Chen H, Sandler DP, Taylor JA, Shore DL, Liu E, Bloomfield CD, Bell DA. Increased risk for myelodysplastic syndromes in individuals with glutathione transferase theta 1 (GSTT1) gene defect. Lancet. 1996 Feb 3;347(8997):295-7. doi: 10.1016/s0140-6736(96)90468-7. PMID 8569364
- [Result] Heinonen K, Mrózek K, Lawrence D, et al.: Trisomy 11 as the sole karyotypic abnormality identifies a group of older patients with acute myeloid leukemia (AML) with FAB M2 or M1 and unfavorable clinical outcome. Results of CALGB 8461. [Abstract] Proc Am Assoc Cancer Res 37: A-1275, 186-7, 1996.
- [Result] Slack JL, Arthur DC, Lawrence D, Mrozek K, Mayer RJ, Davey FR, Tantravahi R, Pettenati MJ, Bigner S, Carroll AJ, Rao KW, Schiffer CA, Bloomfield CD. Secondary cytogenetic changes in acute promyelocytic leukemia--prognostic importance in patients treated with chemotherapy alone and association with the intron 3 breakpoint of the PML gene: a Cancer and Leukemia Group B study. J Clin Oncol. 1997 May;15(5):1786-95. doi: 10.1200/JCO.1997.15.5.1786. PMID 9164186
- [Derived] Archer KJ, Fu H, Mrozek K, Nicolet D, Mims AS, Uy GL, Stock W, Byrd JC, Hiddemann W, Braess J, Spiekermann K, Metzeler KH, Herold T, Eisfeld AK. Identifying long-term survivors and those at higher or lower risk of relapse among patients with cytogenetically normal acute myeloid leukemia using a high-dimensional mixture cure model. J Hematol Oncol. 2024 May 3;17(1):28. doi: 10.1186/s13045-024-01553-6. PMID 38702786
- [Derived] Ozga M, Nicolet D, Mrozek K, Yilmaz AS, Kohlschmidt J, Larkin KT, Blachly JS, Oakes CC, Buss J, Walker CJ, Orwick S, Jurinovic V, Rothenberg-Thurley M, Dufour A, Schneider S, Sauerland MC, Gorlich D, Krug U, Berdel WE, Woermann BJ, Hiddemann W, Braess J, Subklewe M, Spiekermann K, Carroll AJ, Blum WG, Powell BL, Kolitz JE, Moore JO, Mayer RJ, Larson RA, Uy GL, Stock W, Metzeler KH, Grimes HL, Byrd JC, Salomonis N, Herold T, Mims AS, Eisfeld AK. Sex-associated differences in frequencies and prognostic impact of recurrent genetic alterations in adult acute myeloid leukemia (Alliance, AMLCG). Leukemia. 2024 Jan;38(1):45-57. doi: 10.1038/s41375-023-02068-8. Epub 2023 Nov 28. PMID 38017103
- [Derived] Rebechi M, Kohlschmidt J, Mrozek K, Nicolet D, Mims AS, Blachly JS, Orwick S, Larkin KT, Oakes CC, Hantel A, Carroll AJ, Blum WG, Powell BL, Uy GL, Stone RM, Larson RA, Byrd JC, Paskett ED, Plascak JJ, Eisfeld AK. Association of social deprivation with survival in younger adult patients with AML: an Alliance study. Blood Adv. 2023 Aug 8;7(15):4019-4023. doi: 10.1182/bloodadvances.2022009325. No abstract available. PMID 37196637
- [Derived] Mrozek K, Kohlschmidt J, Blachly JS, Nicolet D, Carroll AJ, Archer KJ, Mims AS, Larkin KT, Orwick S, Oakes CC, Kolitz JE, Powell BL, Blum WG, Marcucci G, Baer MR, Uy GL, Stock W, Byrd JC, Eisfeld AK. Outcome prediction by the 2022 European LeukemiaNet genetic-risk classification for adults with acute myeloid leukemia: an Alliance study. Leukemia. 2023 Apr;37(4):788-798. doi: 10.1038/s41375-023-01846-8. Epub 2023 Feb 23. PMID 36823396
- [Derived] Fobare S, Kohlschmidt J, Ozer HG, Mrozek K, Nicolet D, Mims AS, Garzon R, Blachly JS, Orwick S, Carroll AJ, Stone RM, Wang ES, Kolitz JE, Powell BL, Oakes CC, Eisfeld AK, Hertlein E, Byrd JC. Molecular, clinical, and prognostic implications of PTPN11 mutations in acute myeloid leukemia. Blood Adv. 2022 Mar 8;6(5):1371-1380. doi: 10.1182/bloodadvances.2021006242. PMID 34847232
- [Derived] Mims AS, Kohlschmidt J, Borate U, Blachly JS, Orwick S, Eisfeld AK, Papaioannou D, Nicolet D, Mromicronzek K, Stein E, Bhatnagar B, Stone RM, Kolitz JE, Wang ES, Powell BL, Burd A, Levine RL, Druker BJ, Bloomfield CD, Byrd JC. A precision medicine classification for treatment of acute myeloid leukemia in older patients. J Hematol Oncol. 2021 Jun 23;14(1):96. doi: 10.1186/s13045-021-01110-5. PMID 34162404
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516
- [Derived] Niederwieser C, Nicolet D, Carroll AJ, Kolitz JE, Powell BL, Kohlschmidt J, Stone RM, Byrd JC, Mrozek K, Bloomfield CD. Chromosome abnormalities at onset of complete remission are associated with worse outcome in patients with acute myeloid leukemia and an abnormal karyotype at diagnosis: CALGB 8461 (Alliance). Haematologica. 2016 Dec;101(12):1516-1523. doi: 10.3324/haematol.2016.149542. Epub 2016 Jul 28. PMID 27470602